CLINICAL TRIAL: NCT01015144
Title: The Influence of Atorvastatin on the Parameters of Inflammation and the Function of Left Ventricle in Patients With Dilated Cardiomyopathy
Brief Title: The Influence of Atorvastatin on the Parameters of Inflammation and the Function of Left Ventricle
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Agata Bielecka-Dąbrowa, UM Lodz
Other Study IDs: 502-11-585
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Dilated Cardiomyopathy
Keywords: atorvastatin; dilated cardiomyopathy; heart failure; inflammation
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure; Inflammation | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood68
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Atorvastatin
  Interventions: Drug: Tulip
- No statin

INTERVENTIONS:
Drug: Tulip — Patients were divided into two groups: A, who were administered atorvastatin 40 mg daily for two months and 10 mg for next 4 months; and group B, 4 who were treated according to current guidelines without statin therapy.
  Groups: Atorvastatin

SUMMARY:
The aim of the study was to assess of the influence of atorvastatin on selected indicators of an inflammatory condition, function of the left ventricle and factors affecting the occurrence of undesired events like rehospitalizations and mortality in patients with dilated cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years old or older
* patients who signed informed consent
* patients with dilated cardiomyopathy (according ESC 2007)
* patients who had no significant coronary artery stenoses >30% on cardiac catheterization

Exclusion Criteria:

* BP ≥140/90 lub <90/60
* congenital heart disease
* acquired valvular disease except for mitral incompetence secondary to left ventricular dilatation
* New York Heart Association (NYHA) functional class IV
* statin treatment
* preserved hyperactivity of aminotransferases with unexplained etiology,
* muscle disorders which might cause drug-induced myopathy,
* uncontrolled diabetes,
* liver diseases,
* creatinine level > 2 mg/dl and/or GFR<30ml/min,
* abuse of alcohol or drugs,
* chronic inflammatory diseases,
* pregnancy or lactation,
* severe hypothyroidism,
* immunosuppressive treatment,
* operation or severe injury during last month
* vaccination during last 3 months
* heart stimulation device or implantable cardioverter defibrillator
* or who didn't write conscious consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dilated cardiomyopathy (according ESC 2007) with EF≤40% as documented by echocardiography were included.
Sampling Method: Probability Sample
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
left ventricular function | 2 months

SECONDARY OUTCOMES:
mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Agata Bielecka-Dabrowa, PhD, Principal Investigator — Department of Hypertension UM Lodz; Maciej Banach, Assoc. Prof., Study Director — Department of Hypertension UM Lodz

REFERENCES:
- [Background] Bielecka-Dabrowa A, Wierzbicka M, Dabrowa M, Goch A. New methods in laboratory diagnostics of dilated cardiomyopathy. Cardiol J. 2008;15(4):388-95. PMID 18698552
- [Background] Bielecka-Dabrowa A, Wierzbicka M, Goch JH. [Proinflammatory cytokines in cardiovascular diseases as potential therapeutic target]. Wiad Lek. 2007;60(9-10):433-8. Polish. PMID 18350717
- [Derived] Bielecka-Dabrowa A, Goch JH, Rysz J, Maciejewski M, Desai R, Aronow WS, Banach M. Influence of co-existing atrial fibrillation on the efficacy of atorvastatin treatment in patients with dilated cardiomyopathy: a pilot study. Lipids Health Dis. 2010 Feb 23;9:21. doi: 10.1186/1476-511X-9-21. PMID 20178563
- [Derived] Bielecka-Dabrowa A, Goch JH, Mikhailidis DP, Rysz J, Maciejewski M, Banach M. The influence of atorvastatin on parameters of inflammation and function of the left ventricle in patients with dilated cardiomyopathy. Med Sci Monit. 2009 Dec;15(12):MS12-23. PMID 19946241